CLINICAL TRIAL: NCT01809353
Title: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Crossover Study to Evaluate the Pharmacokinetics and Safety of JNJ-54452840 Following Single Intravenous Doses to Healthy Japanese and Caucasian Subjects
Brief Title: To Assess the Pharmacokinetics and Safety of Single Doses of JNJ-54452840 in Healthy Japanese and Caucasian Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Janssen Research & Development, LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: CR100982; 54452840HFA1001 (Other: Janssen Research & Development, LLC)
Record Dates: First submitted 2013-03-08; First posted 2013-03-12 (Estimated); Last update posted 2015-03-23 (Estimated); Status verified 2015-03

CONDITIONS: Healthy
Keywords: Healthy; Japanese; Caucasian; Male; Pharmacokinetic; JNJ-54452840
MeSH Terms: interventions — JNJ-54452840

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (8):
- Group A: JNJ-54452840 20 mg (Experimental): Each participant will receive 20 mg of JNJ-54452840 as a single intravenous dose.
  Interventions: Drug: JNJ-54452840
- Group A: JNJ-54452840 80 mg (Experimental): Each participant will receive 80 mg of JNJ-54452840 as a single intravenous dose.
  Interventions: Drug: JNJ-54452840
- Group A: JNJ-54452840 240 mg (Experimental): Each participant will receive 240 mg of JNJ-54452840 as a single intravenous dose.
  Interventions: Drug: JNJ-54452840
- Group A: Placebo (Placebo Comparator): Each participant will receive matching placebo as a single intravenous dose.
  Interventions: Other: Placebo
- Group B: JNJ-54452840 20 mg (Experimental): Each participant will receive 20 mg of JNJ-54452840 as a single intravenous dose.
  Interventions: Drug: JNJ-54452840
- Group B: JNJ-54452840 80 mg (Experimental): Each participant will receive 80 mg of JNJ-54452840 as a single intravenous dose.
  Interventions: Drug: JNJ-54452840
- Group B: JNJ-54452840 240 mg (Experimental): Each participant will receive 240 mg of JNJ-54452840 as a single intravenous dose.
  Interventions: Drug: JNJ-54452840
- Group B: Placebo (Placebo Comparator): Each participant will receive matching placebo as a single intravenous dose.
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: JNJ-54452840 — Single intravenous (medication is injected into a vein) doses of 20 mg, 80 mg, and 240 mg
  Arms: Group A: JNJ-54452840 20 mg; Group A: JNJ-54452840 240 mg; Group A: JNJ-54452840 80 mg; Group B: JNJ-54452840 20 mg; Group B: JNJ-54452840 240 mg; Group B: JNJ-54452840 80 mg
Other: Placebo — Single matching intravenous dose
  Arms: Group A: Placebo; Group B: Placebo

SUMMARY:
The purpose of this study is to assess the pharmacokinetics (ie, how the body affects the drug) and safety of JNJ-54452840 in healthy participants.

DETAILED DESCRIPTION:
This is a Phase 1, randomized (the study treatment is assigned by chance), double-blind (neither physician nor participant knows the treatment received), placebo-controlled (one of the study treatments is inactive), four-way cross-over study (method used to switch participants from one treatment arm to another in a clinical trial) conducted in healthy male Japanese and Caucasian participants. The study will be conducted in 3 parts; a screening phase (up to 28 days), a double-blind treatment phase (28 days), and a follow-up phase (approximately 21 to 28 days). The study will be conducted in 2 groups (Group A consists of 16 Japanese participants; Group B consists of 16 Caucasian participants) over 4 treatment periods. On Day 1 of Period 1, approximately 16 eligible Japanese participants and the same number of eligible Caucasian participants will be randomly assigned to 1 of 4 treatment sequences and will receive the 4 intravenous treatments JNJ-54452840 20 mg, JNJ-54452840 80 mg, JNJ-54452840 240 mg, and placebo across the treatment periods according to the order specified by the randomization schedule.

Participants will come to the study center each time they receive study medication and will be discharged from the study center 24 hours after dosing during each treatment period after satisfactory review of all clinical safety measures. Blood samples will be drawn at time points during the treatment and follow-up periods for participants in both Group A and Group B of the study. Participants will return to the study center for a follow-up visit within approximately 7 to 10 days after the last study procedure in the last treatment period for safety assessments, followed by another visit within approximately 21 to 28 days for assessment of anti -beta-1-AR (adrenergic receptor) auto-antibodies in blood (auto-antibodies targeting the human beta-1-AR antibody). If anti-beta-1-AR auto-antibodies are detected at this second follow-up visit, additional testing will be performed every 3 months until autoantibody levels fall below the level of detection of the assay or for 1 year, whichever occurs earlier. Participants in Group A and Group B will be involved in the study for approximately 12 weeks and up to 1 year if they develop anti -beta-1-AR auto-antibodies . Safety of the participants will be monitored throughout the study.

ELIGIBILITY:
Inclusion Criteria:

* Must be a healthy male with no clinically relevant abnormalities as determined by medical history, physical examination, blood chemistry assessments, hematologic assessments - Must be Japanese or Caucasian
* Japanese participants must have been born in Japan, have resided outside of Japan for no more than 5 years, and have Japanese parents and maternal and paternal grandparents
* Caucasian participants must have Caucasian parents

Exclusion Criteria:

* History of or current clinically significant medical illness that the investigator considers should exclude the participant or that could interfere with the interpretation of the study results
* Have a known or suspected intolerance or hypersensitivity to any biologic medication or known allergies or clinically significant reactions to murine, chimeric, or human peptides or protein
* Be unable or unwilling to undergo multiple venipunctures because of poor tolerability or lack of easy access to veins

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 32 (Actual)
Dates: Start 2013-07; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Serum concentrations of JNJ-54452840 | Up to Day 2
  Serum concentrations of JNJ-54452840 will be used to determine pharmacokinetic parameters for JNJ-54452840

SECONDARY OUTCOMES:
Number of participants with an adverse event as a measure of safety | Up to Day 2

CONTACTS AND LOCATIONS:
Overall Officials: Janssen Research & Development, LLC Clinical Trial, Study Director — Janssen Research & Development, LLC
Locations (1):
- Cypress, California, United States

REFERENCES:
- See also: A Phase 1 Randomized, Double-Blind, Placebo-Controlled Crossover Study to Evaluate the Pharmacokinetics and Safety of JNJ-54452840 Following Single Intravenous Doses to Healthy Male Japanese and Caucasian Subjects — http://filehosting.pharmacm.com/DownloadService.ashx?client=CTR_JNJ_6051&studyid=3650&filename=CR100982_CSR.pdf